CLINICAL TRIAL: NCT01949116
Title: Effect of Reducing Inflammation With Low Dose Methotrexate on Inflammatory Markers and Endothelial Function in Treated and Suppressed HIV Infection
Brief Title: Safety and Effectiveness of Low-Dose Methotrexate for Reducing Inflammation in HIV-Infected Adults on ARV Medications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A5314; 11875 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-dose methotrexate (LDMTX) (Experimental): From study entry through Week 1, participants received 5 mg of LDMTX once a week. For participants who were clinically stable at the Week 1 study visit, the dose of LDMTX was increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose of LDMTX was increased to 15 mg once a week through Week 24. Participants who did not meet the criteria for dose escalation were re-evaluated at the following study visit. In addition to LDMTX, all participants also received 1 mg of folic acid once a day from study entry throughout Week 24. After taking the final dose of LDMTX, all participants continued taking folic acid for an additional 4 weeks.
  Interventions: Drug: LDMTX; Dietary Supplement: Folic acid
- Placebo (Placebo Comparator): From study entry through Week 1, participants received 5 mg of placebo once a week. For participants who were clinically stable at the Week 1 study visit, the dose of placebo was increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose of placebo was increased to 15 mg once a week through Week 24. Participants who did not meet the criteria for dose escalation were re-evaluated at the following study visit. In addition to placebo, all participants also received 1 mg of folic acid once a day from study entry throughout Week 24. After taking the final dose of placebo, all participants continued taking folic acid for an additional 4 weeks.
  Interventions: Drug: Placebo; Dietary Supplement: Folic acid

INTERVENTIONS:
Drug: LDMTX — LDMTX 5 mg: one 5-mg capsule by mouth once weekly
  LDMTX 10 mg: two 5-mg capsules by mouth once weekly
  LDMTX 15 mg: three 5-mg capsules by mouth once weekly
  Other Names: Low-Dose Methotrexate
  Arms: Low-dose methotrexate (LDMTX)
Drug: Placebo — Placebo 5 mg: one 5-mg capsule by mouth once weekly
  Placebo 10 mg: two 5-mg capsules by mouth once weekly
  Placebo 15 mg: three 5-mg capsules by mouth once weekly
  Other Names: Placebo for Low-Dose Methotrexate
  Arms: Placebo
Dietary Supplement: Folic acid — 1-mg tablet of folic acid by mouth once a day

SUMMARY:
People with HIV infection who are taking antiretroviral therapy (ART) could be at risk for cardiovascular disease (CVD), which can be caused by inflammation. Methotrexate (MTX) is a medication used to treat inflammation in people with rheumatoid arthritis. This study evaluated the safety and effectiveness of low-dose methotrexate (LDMTX) at reducing inflammation in HIV-infected adults.

DETAILED DESCRIPTION:
HIV-infected people taking ART have a higher than expected risk of premature CVD. Many factors likely contribute to this risk, including chronic inflammation. Strategies to reduce inflammation in HIV-infected people may be beneficial in reducing CVD risk, as well as other conditions, including kidney disease, bone disease, and neurologic complications. MTX is an anti-inflammatory medication used to treat people with rheumatoid arthritis. This study evaluated the safety and effectiveness of LDMTX at treating inflammation and on endothelial function in virologically suppressed HIV-infected adults who had CVD or were at increased risk of CVD.

The total study duration was 36 weeks. Prior to enrolling in the study, participants had a chest X-ray. Participants were randomly assigned to receive LDMTX or placebo for 24 weeks. Participants continued taking their antiretroviral (ARV) medications as usual; ARVs were not provided by the study. At study entry, participants underwent a medical and medication history, physical examination, blood collection, and adherence assessments. From study entry through Week 1, participants received either 5 mg of LDMTX or placebo once a week. For participants who were clinically stable at the Week 1 study visit, the dose of LDMTX or placebo was increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose of LDMTX or placebo was increased to 15 mg once a week through Week 24. Participants who did not meet the criteria for dose escalation were re-evaluated at the following study visit. In addition to LDMTX or placebo, all participants also received 1 mg of folic acid once a day from study entry throughout Week 24. After taking the final dose of LDMTX or placebo, all participants continued taking folic acid for an additional 4 weeks.

Post-entry visits occurred at Weeks 1, 2, 4, 8, 12, 18, 24, and 36. These included a physical examination, blood collection, and adherence assessments; an arm ultrasound test was performed at Weeks 12 and 24. At Week 2, some participants took part in a pharmacokinetic (PK) assessment, which involved undergoing a blood collection several times over a 6-hour period.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.
* Had to be on continuous ART for greater than or equal to 24 weeks prior to study entry. This was defined as continuous active therapy for the 24-week period prior to study entry with no treatment interruption longer than 7 consecutive days and a total duration off treatment of no more than 14 days in the 90 days prior to study entry.
* CD4 T-cell count greater than or equal to 400 cells/mm^3 obtained within 60 days prior to study entry by any U.S. laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent
* HIV-1 RNA level below the limit of quantification using a FDA-approved assay for at least 24 weeks prior to study entry and confirmed within 60 days prior to study entry. The assay used for eligibility could be performed by any U.S. laboratory that had a CLIA certification or its equivalent. NOTE: Single determinations that are between the assay quantification limit and 200 copies/mL were allowed as long as the preceding and subsequent determinations are below the level of quantification.
* The following laboratory values obtained within 60 days prior to study entry by any U.S. laboratory that has a CLIA certification or its equivalent:

  1. Fasting glucose less than 180 mg/dL
  2. Alanine aminotransferase (ALT) [serum glutamic pyruvic transaminase (SGPT)] less than 2 times the upper limit of normal (ULN)
  3. Aspartate aminotransferase (AST) [serum glutamic oxaloacetic transaminase (SGOT)] less than 2 times the ULN
  4. Estimated creatinine clearance (CrCl) greater than or equal to 50 mL/min by Cockcroft-Gault. NOTE: Candidates who were taking tenofovir disoproxil fumarate (TDF) as part of their ART regimen should have an estimated CrCl greater than or equal to 60 mL/min.
  5. White blood cell (WBC) greater than 3,000/mm^3
  6. Hemoglobin greater than 12.0 g/dL
  7. Platelets greater than 150,000/mm^3
* Female candidates who were postmenopausal (i.e., of non-childbearing potential) were defined as having either:

  1. Appropriate medical documentation of prior hysterectomy and/or complete bilateral oophorectomy (i.e., surgical removal of the ovaries, resulting in "surgical menopause" and occurring at the age at which the procedure was performed), OR
  2. Permanent cessation of previously occurring menses as a result of ovarian failure with documentation of hormonal deficiency by a certified healthcare provider (i.e., "spontaneous menopause").
* Male candidates must agree not to participate in a conception process (i.e., active attempt to impregnate, sperm donation). If participating in sexual activity that could lead to pregnancy, the male participant must agree to the use of TWO reliable forms of contraceptives simultaneously while on study and for a minimum of 3 months after therapy.
* Candidates who were not of reproductive potential (defined as women who have been postmenopausal for at least 24 consecutive months or men who have documented vasectomy) were eligible for the study without requiring the use of contraceptives.
* Moderate or high CVD risk defined as:

A) Documented CVD as assessed by meeting at least 1 of 3 criteria below:

1. Coronary artery disease (CAD): prior myocardial infarction (MI) due to atherosclerosis, coronary artery bypass graft surgery, percutaneous coronary intervention, or angiographic CAD with luminal diameter stenosis of at least one coronary artery at least 50%.
2. Cerebrovascular disease: prior ischemic stroke of carotid origin, carotid endarterectomy or stenting, or angiographic carotid stenosis of at least 50%.
3. Peripheral arterial disease: prior lower extremity arterial surgical or percutaneous revascularization procedure, or angiographic lower extremity arterial stenosis of at least 50%.

OR

B) Controlled type II diabetes mellitus (HbA1C less than or equal to 8.0% within the past 90 days prior to study entry, regardless of use of medications)

OR

C) Any one of the following CVD risk factors below:

1. Current smoking: self-report of smoking at least a half a pack of cigarettes a day, on average, in the past month.
2. Hypertension (HTN): two consecutive blood pressure (BP) readings with either systolic greater than 140 mm Hg or diastolic greater than 90 mm Hg; or on antihypertensive medications.
3. Dyslipidemia: defined as non-high-density lipoprotein (HDL)-C greater than 160 mg/dL or HDL-C less than or equal to 40 mg/dL, regardless of medication use.
4. High-sensitivity C-reactive protein (hsCRP) greater than or equal to 2 mg/L at screening

Ability and willingness of candidate to provide informed consent

* Completion of the Flow-mediated Vasodilation (FMD) assessments. NOTE: The FMD must be performed at the site and confirmed as acceptable by the University of Wisconsin Atherosclerosis Imaging Research Program (UW AIRP) core lab prior to study entry. If the FMD is deemed unacceptable, a repeat scan must be performed prior to enrollment.
* Appropriate documentation from medical records of prior receipt of pneumococcal vaccination (with both the 13-valent conjugant vaccine [PCV13] and 23-valent pneumococcal polysaccharide vaccine [PPV23]) within the last 5 years. If no documentation is available, then the PCV13 and PPV23 series (PCV13 vaccine followed by PPV23 vaccine at least 8 weeks later) should be completed more than 14 days prior to study entry.

Exclusion Criteria:

* Acute or serious illness requiring systemic treatment and/or hospitalization within 60 days prior to study entry. NOTE: Treatment should have ended at least 60 days prior to study entry for eligibility.
* Documentation of any CDC category C AIDS-indicator condition or oropharyngeal candidiasis (thrush) within 90 days prior to study entry
* Receipt of antibiotic therapy within 30 days prior to study entry
* Latent tuberculosis (TB) infection (defined as a positive purified protein derivative [PPD] greater than or equal to 5 mm, positive interferon-gamma release assay, or positive T-spot test at any time in the past) or evidence of latent TB on the screening chest x-ray that had not been completely treated or was treated within the past 6 months prior to study entry
* TB disease that required treatment within 48 weeks prior to study entry
* Life-threatening fungal infection requiring treatment, in the opinion of the site investigator, within 48 weeks prior to study entry
* Herpes-zoster viral infection that required treatment within 90 days prior to study entry
* A history of or current, active hepatitis B infection defined as positive hepatitis B surface antigen (HBsAg) test or positive hepatitis B virus (HBV) DNA in candidates with isolated hepatitis B core antibody (HBcAb) positivity, defined as negative HBsAg, negative hepatitis B surface antibody (HBsAb), and positive HBcAb within 24 weeks prior to study entry. NOTE: Candidates who were positive for hepatitis B surface antigen but who were HBV DNA negative were permitted in the study.
* Chronic hepatitis C infection defined as a positive hepatitis C antibody and positive hepatitis C RNA at any time prior to study entry. NOTE: Candidates who were positive for hepatitis C antibody but whowerehepatitis C virus (HCV) RNA negative are permitted in the study. Candidates who had been treated for hepatitis C should be HCV RNA negative for at least 24 weeks after completion of therapy to be eligible for the study.
* Previously diagnosed myelodysplasia syndrome
* Treated lymphoproliferative disease less than or equal to 5 years prior to study entry
* Clinically significant lung disease on the screening chest x-ray that, in the opinion of the site investigator, places the candidate at increased risk of lung toxicity (e.g., history of pulmonary fibrosis, interstitial lung disease, or pulmonary lymphoproliferative disease)
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry
* Change in the ART regimen in the 12 weeks prior to study entry or intended modification of ART during the study. NOTE: Modifications of ART doses during the 12 weeks prior to study entry were permitted. In addition, the change in formulation (e.g., from standard formulation to fixed-dose combination) was allowed within 12 weeks prior to study entry. A within class single drug substitution (e.g., switch from nevirapine to efavirenz or from atazanavir to darunavir) is allowed within 12 weeks prior to study entry, with the exception of a switch from any other nucleoside reverse transcriptase inhibitor (NRTI) to abacavir. No other changes in ART in the 12 weeks prior to study entry were permitted.
* Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation
* Average daily consumption of three or more alcoholic beverages for 4 weeks prior to study entry or intention to consume an average of two or more alcoholic beverages a day during the study. NOTE: An alcohol-containing beverage is defined as 12 ounces of beer, 4 ounces of wine, or 1 ounce of spirits.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Changes in lipid-lowering or antihypertensive medication within 90 days prior to study entry or expected need to modify these medications during the study. NOTE: Lipid-lowering medication includes: statins, fibrates, niacin (dose greater than or equal to 250 mg daily), and fish-oil/omega 3 fatty acids (dose greater than 1000 mg of marine oils daily).
* Vaccination (e.g., influenza, pneumococcal polysaccharide) within 14 days prior to study entry
* Anticipated need to receive vaccination (e.g., influenza, pneumococcal polysaccharide) within 1 week prior to Week 4, 12, 24, or 36 study visits
* Excess extracompartmental fluids including ascites, pericardial fluid, and pleural effusions which, in the opinion of the study investigators, would result in difficulty in monitoring the dose of MTX
* Use of drugs that alter folic acid metabolism such as trimethoprim/sulfamethoxazole or reduce tubular excretion such as probenecid within 14 days prior to study entry
* New York Heart Association Class IV congestive heart failure
* Diabetes mellitus with HbA1C greater than 8.0% within the past 90 days prior to study entry

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2016-12-08 (Actual); Study Completion 2016-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Hsue, MD, Study Chair — San Francisco General Hospital; Judith Currier, MD, MSc, Study Chair — University of California, Los Angeles
Locations (22):
- United States (22):
  - Alabama CRS, Birmingham, Alabama
  - University of Southern California CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - Harbor-UCLA CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Brigham and Women's Hospital Therapeutics Clinical Research Site (BWH TCRS) CRS, Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Greensboro CRS, Greensboro, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Case Clinical Research Site, Cleveland, Ohio
  - Ohio State University CRS, Columbus, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - Houston AIDS Research Team CRS, Houston, Texas

REFERENCES:
- [Derived] Cyktor JC, Yeh E, Ribaudo H, Hoeth D, Naqvi A, Bell T, Ridker PM, Fichtenbaum C, Daar ES, Havlir D, Tawakol A, Lederman MM, Stein JH, Deeks SG, Currier JS, Hsue PY, Mellors JW; A5314 Team. Brief Report: Low-Dose Methotrexate Does Not Affect Measures of HIV-1 Persistence in Individuals With Chronically Treated HIV-1 Infection. J Acquir Immune Defic Syndr. 2024 Aug 15;96(5):481-485. doi: 10.1097/QAI.0000000000003453. PMID 39287554
- [Derived] Hsue PY, Ribaudo HJ, Deeks SG, Bell T, Ridker PM, Fichtenbaum C, Daar ES, Havlir D, Yeh E, Tawakol A, Lederman M, Currier JS, Stein JH. Safety and Impact of Low-dose Methotrexate on Endothelial Function and Inflammation in Individuals With Treated Human Immunodeficiency Virus: AIDS Clinical Trials Group Study A5314. Clin Infect Dis. 2019 May 17;68(11):1877-1886. doi: 10.1093/cid/ciy781. PMID 30219823
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification, August 2009) — http://rsc.tech-res.com/safetyandpharmacovigilance/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 176 participants randomized to A5314 - 86 in LDMTX, 90 in Placebo. The first participant enrolled on January 31, 2014; the last participant enrolled on March 31, 2016. A range of 2 to 25 participants per site enrolled across 22 clinical research sites during study accrual.
Groups:
- Low-dose Methotrexate (LDMTX): From study entry through Week 1, participants received 5 mg of LDMTX once a week. For participants who were clinically stable at the Week 1 study visit, the dose of LDMTX was increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose of LDMTX was increased to 15 mg once a week through Week 24. Participants who did not meet the criteria for dose escalation were re-evaluated at the following study visit. In addition to LDMTX, all participants also received 1 mg of folic acid once a day from study entry throughout Week 24. After taking the final dose of LDMTX, all participants continued taking folic acid for an additional 4 weeks.
  LDMTX: LDMTX 5 mg: one 5-mg capsule by mouth once weekly
  LDMTX 10 mg: two 5-mg capsules by mouth once weekly
  LDMTX 15 mg: three 5-mg capsules by mouth once weekly
  Folic acid: 1-mg tablet of folic acid by mouth once a day
- Placebo: From study entry through Week 1, participants received 5 mg of placebo once a week. For participants who were clinically stable at the Week 1 study visit, the dose of placebo was increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose of placebo was increased to 15 mg once a week through Week 24. Participants who did not meet the criteria for dose escalation were re-evaluated at the following study visit. In addition to placebo, all participants also received 1 mg of folic acid once a day from study entry throughout Week 24. After taking the final dose of placebo, all participants continued taking folic acid for an additional 4 weeks.
  Placebo: Placebo 5 mg: one 5-mg capsule by mouth once weekly
  Placebo 10 mg: two 5-mg capsules by mouth once weekly
  Placebo 15 mg: three 5-mg capsules by mouth once weekly
  Folic acid: 1-mg tablet of folic acid by mouth once a day
Period: Overall Study
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Started | 86 | 90
Completed | 78 | 84
Not Completed | 8 | 6
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population consists of all eligible participants who were randomized for the study.
Groups:
- Low-dose Methotrexate (LDMTX): From study entry through Week 1, participants will receive 5 mg of LDMTX once a week. For participants who are clinically stable at the Week 1 study visit, the dose will be increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose will be increased to 15 mg once a week through Week 24. In addition to LDMTX, all participants will also receive 1 mg of folic acid once a day from study entry through 4 weeks after LDMTX is discontinued, either at Week 24 or earlier, for any reason.
  LDMTX: LDMTX 5 mg: one 5-mg capsule by mouth once weekly
  LDMTX 10 mg: two 5-mg capsules by mouth once weekly
  LDMTX 15 mg: three 5-mg capsules by mouth once weekly
  Folic acid: 1-mg tablet of folic acid by mouth once a day
- Placebo: From study entry through Week 1, participants will receive 5 mg of placebo once a week. For participants who are clinically stable at the Week 1 study visit, the dose will be increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose will be increased to 15 mg once a week through Week 24. In addition to placebo, all participants will also receive 1 mg of folic acid once a day from study entry through 4 weeks after placebo is discontinued, either at Week 24 or earlier, for any reason.
  Placebo: Placebo 5 mg: one 5-mg capsule by mouth once weekly
  Placebo 10 mg: two 5-mg capsules by mouth once weekly
  Placebo 15 mg: three 5-mg capsules by mouth once weekly
  Folic acid: 1-mg tablet of folic acid by mouth once a day
- Total: Total of all reporting groups
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo | Total
Number analyzed (Participants) | 86 | 90 | 176
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [51 to 60] | 53 [49 to 56] | 54 [49 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 78 | 81 | 159
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 86 | 90 | 176
Current Statin Use [Count of Participants; unit: Participants] — Current Statin Use at Study Entry - this is a stratification factor for the study.
  Participants
    Current Statin Use | 51 | 52 | 103
    No Current Statin Use | 35 | 38 | 73
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 28 | 40 | 68
  Current non-smoker | 58 | 50 | 108
Type of CVD Risk [Count of Participants; unit: Participants] — CVD = cardiovascular disease; CAD = coronary artery disease; PAD = peripheral artery disease; hsCRP = high-sensitivity C-reactive protein.
  Participants
    CAD, CVD, or PAD | 20 | 12 | 32
    Controlled type 2 diabetes mellitus | 19 | 20 | 39
    Smoking/hypertension/dyslipidemia/hsCRP >= 2mg/L | 47 | 58 | 105
10 year ASCVD risk [Median (Inter-Quartile Range); unit: Percent risk of ASCVD] — Atherosclerotic cardiovascular disease (ASCVD) is defined as coronary death or nonfatal myocardial infarction, or fatal or nonfatal stroke, based on the Pooled Cohort Equations. The 10-year risk was calculated for only those participants who fell in the CVD Risk category, "Smoking, hypertension, dyslipidemia, or hsCRP >= 2 mg/L." Population: Participants with any risk of CAD, CVD, PAD, or controlled type 2 diabetes mellitus are excluded from the ASCVD risk calculation.
  Percent risk of ASCVD
    number analyzed (Participants) | 47 | 58 | 105
    (all) | 10.1 [5.4 to 14.3] | 7.9 [5.0 to 12.4] | 8.7 [5.1 to 13.0]
CD4+ cell count [Median (Inter-Quartile Range); unit: cells/mm^3] | 689 [551 to 910] | 729 [569 to 947] | 726 [552 to 940]
HIV-1 RNA [Count of Participants; unit: Participants]
  Detectable | 2 | 4 | 6
  Below Assay Limit of Detection | 84 | 84 | 168
  Missing | 0 | 2 | 2
Brachial Artery FMD [Median (Inter-Quartile Range); unit: Percent Dilation] — Flow-mediated vasodilation is defined as the maximum FMD (%) calculated from reactive hyperemia (RH) 60 and RH 90 relative to resting artery diameter. Population: 3 participants in the placebo group have either unsatisfactory scans or did not meet protocol requirements at the time of the FMD assessment.
  Percent Dilation
    number analyzed (Participants) | 86 | 87 | 173
    (all) | 3.54 [2.19 to 4.91] | 3.41 [1.98 to 5.03] | 3.45 [2.10 to 4.91]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reached at Least One Safety Milestone Over the Duration of Study Follow-up (36 Weeks)
Description: Number of participants who experienced any one of the following safety milestones:
  * Entry CD4+ T-cell count less than 700 cells/mm^3, confirmed CD4+ decline greater than 33% of baseline AND to less than 350 cells/mm^3
  * Entry CD4+ T-cell count greater than or equal to 700 cells/mm^3, a confirmed CD4+ decline greater than 50% of baseline
  * Confirmed HIV-1 RNA Level Greater Than 200 Copies/mL in the Absence of an Interruption in ART
  * New or recurrent CDC category C AIDS-indicator condition
  * Evidence of HIV-associated infection including CMV end-organ disease, varicella zoster, EBV related clinical disease
  * Requirement for LDMTX discontinuation for confirmed Grade 3 or higher toxicity
  * Lymphoproliferative malignancies
  * Pulmonary toxicity which is defined as Grade 3 or 4 dyspnea, cough, shortness of breath which in the opinion of the local investigator is related to the study drug but not related to other clinical causes such as asthma, influenza, etc.
Time Frame: From study entry to week 36
Population: Intent-to-treat (ITT) population consists of all eligible participants who were randomized for the study.
Measure: Count of Participants; unit: Participants
Groups:
- Low-dose Methotrexate (LDMTX): From study entry through Week 1, participants will receive 5 mg of LDMTX once a week. For participants who are clinically stable at the Week 1 study visit, the dose will be increased to 10 mg once a week through Week 12. For participants who are clinically stable at the Week 12 study visit, the dose will be increased to 15 mg once a week through Week 24. In addition to LDMTX, all participants will also receive 1 mg of folic acid once a day from study entry through 4 weeks after LDMTX is discontinued, either at Week 24 or earlier, for any reason.
  LDMTX: LDMTX 5 mg: one 5-mg capsule by mouth once weekly
  LDMTX 10 mg: two 5-mg capsules by mouth once weekly
  LDMTX 15 mg: three 5-mg capsules by mouth once weekly
  Folic acid: 1-mg tablet of folic acid by mouth once a day
- Placebo: From study entry through Week 1, participants will receive 5 mg of placebo once a week. For participants who are clinically stable at the Week 1 study visit, the dose will be increased to 10 mg once a week through Week 12. For participants who are clinically stable at the Week 12 study visit, the dose will be increased to 15 mg once a week through Week 24. In addition to placebo, all participants will also receive 1 mg of folic acid once a day from study entry through 4 weeks after placebo is discontinued, either at Week 24 or earlier, for any reason.
  Placebo: Placebo 5 mg: one 5-mg capsule by mouth once weekly
  Placebo 10 mg: two 5-mg capsules by mouth once weekly
  Placebo 15 mg: three 5-mg capsules by mouth once weekly
  Folic acid: 1-mg tablet of folic acid by mouth once a day
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 86 | 90
Participants | 11 | 5
Statistical Analysis 1: Comparison: Low-dose Methotrexate (LDMTX) vs Placebo; Test type: Non-Inferiority — The P-value for the risk difference is from an asymptotic non-inferiority analysis for the proportion (risk) difference with a 15% non-inferiority margin; p = 0.0367, Farrington-Manning score (exact); Risk Difference (RD) = 0.072, 90% CI 1-sided [upper limit 0.134] — LDMTX - Placebo

2. Primary Outcome: Primary Efficacy Endpoint of Change From Baseline to Week 24 in Brachial Artery Flow-mediated Vasodilation (FMD)
Description: Flow-mediated vasodilation is defined as the maximum FMD (%) calculated from reactive hyperemia (RH) 60 and RH 90 relative to resting artery diameter. Absolute change of FMD at week 24 is calculated from baseline FMD.
Time Frame: From Baseline to Week 24
Population: Intent-to-treat (ITT) population consists of all eligible participants who were randomized for the study.
Measure: Mean (95% Confidence Interval); unit: Percent Dilation
Groups:
- Low-dose Methotrexate (LDMTX): From study entry through Week 1, participants received either 5 mg of LDMTX once a week. For participants who were clinically stable at the Week 1 study visit, the dose of LDMTX was increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose of LDMTX was increased to 15 mg once a week through Week 24. Participants who did not meet the criteria for dose escalation was re-evaluated at the following study visit. In addition to LDMTX, all participants also received 1 mg of folic acid once a day from study entry throughout Week 24. After taking the final dose of LDMTX, all participants continued taking folic acid for an additional 4 weeks.
  LDMTX: LDMTX 5 mg: one 5-mg capsule by mouth once weekly
  LDMTX 10 mg: two 5-mg capsules by mouth once weekly
  LDMTX 15 mg: three 5-mg capsules by mouth once weekly
  Folic acid: 1-mg tablet of folic acid by mouth once a day
- Placebo: From study entry through Week 1, participants received either 5 mg of placebo once a week. For participants who were clinically stable at the Week 1 study visit, the dose of placebo was increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose of placebo was increased to 15 mg once a week through Week 24. Participants who did not meet the criteria for dose escalation was re-evaluated at the following study visit. In addition to placebo, all participants also received 1 mg of folic acid once a day from study entry throughout Week 24. After taking the final dose of placebo, all participants continued taking folic acid for an additional 4 weeks.
  Placebo: Placebo 5 mg: one 5-mg capsule by mouth once weekly
  Placebo 10 mg: two 5-mg capsules by mouth once weekly
  Placebo 15 mg: three 5-mg capsules by mouth once weekly
  Folic acid: 1-mg tablet of folic acid by mouth once a day
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 74 | 80
Percent Dilation | 0.24 [-0.40 to 0.88] | 0.15 [-0.47 to 0.77]
Statistical Analysis 1: Comparison: Low-dose Methotrexate (LDMTX) vs Placebo; Test type: Superiority; p = 0.55, Wilcoxon (Mann-Whitney); Stratified by Statin Use (study stratification factor); Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.67 to 0.85]

3. Secondary Outcome: Change From Baseline to Week 12 in Brachial Artery FMD
Description: The absolute change from baseline to week 24 FMD (%), defined as the maximum FMD calculated from reactive hyperemia (RH) 60 and RH 90 relative to resting artery diameter.
Time Frame: From Baseline to Week 12
Population: Intent-to-treat (ITT) population consists of all eligible participants who were randomized for the study.
Measure: Median (Inter-Quartile Range); unit: Percent Dilation
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 74 | 75
Percent Dilation | 0.32 [-1.55 to 1.54] | -0.06 [-1.3 to 1.66]

4. Secondary Outcome: Change From Baseline to Week 12 in Brachial Artery Resting Average Diameter
Description: The change in resting average diameter in millimeters of the brachial artery at week 12 from baseline.
Time Frame: From Baseline to Week 12
Population: Intent-to-treat (ITT) population consists of all eligible participants who were randomized for the study.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 74 | 75
mm | 0.04 [-0.09 to 0.13] | 0.03 [-0.09 to 0.15]

5. Secondary Outcome: Change From Baseline to Week 24 in Brachial Artery Resting Average Diameter
Description: The absolute change in resting average diameter in millimeters of the brachial artery at week 24 from baseline.
Time Frame: From Baseline to Week 24
Population: Intent-to-treat (ITT) population consists of all eligible participants who were randomized for the study.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 74 | 80
mm | 0 [-0.11 to 0.13] | 0.01 [-0.1 to 0.12]

6. Secondary Outcome: Change From Baseline to Week 24 in Reactive Hyperemic (RH) Flow Rate
Description: The absolute change in RH flow rate in cc/min of the brachial artery at week 24 from baseline.
Time Frame: From Baseline to Week 24
Population: Intent-to-treat (ITT) population consists of all eligible participants who were randomized for the study.
Measure: Median (Inter-Quartile Range); unit: cc/min
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 74 | 76
cc/min | -11.40 [-97.46 to 161.64] | 13.76 [-135.11 to 107.73]

7. Secondary Outcome: Change From Baseline to Week 24 in Peak Reactive Hyperemic (RH) Flow Velocity
Description: The absolute change in peak RH flow velocity in cm/s of the brachial artery at week 24 from baseline.
Time Frame: From Baseline to Week 24
Population: Intent-to-treat (ITT) population consists of all eligible participants who were randomized for the study.
Measure: Median (Inter-Quartile Range); unit: cm/s
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 74 | 76
cm/s | -0.20 [-11.30 to 14.40] | -0.83 [-16.80 to 16.88]

8. Secondary Outcome: Percentage Change From Baseline to Week 24 in High-sensitivity C-reactive Protein (hsCRP)
Description: hsCRP is a marker of inflammation. Change from baseline (Week 24 - baseline) was performed on the log10 scale and is thus presented as percentage change, i.e. (10^[fold-change] - 1) x 100%. One single hsCRP result at week 24 was above the limit of quantification, therefore excluded from analysis.
Time Frame: From Baseline to week 24
Population: Adequately-dosed (AD) population included 129 participants who initiated study treatment with 24-week continuous dosing to at least 8 or more 15 mg doses of LDMTX/Placebo (59 in LDMTX, 70 in Placebo). 3 of these participants were not identified at the time of the specimen request for biomarker testing, other missing data are due to missed visits.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Groups:
- Low-dose Methotrexate (LDMTX): From study entry through Week 1, participants received 5 mg of LDMTX once a week. For participants who were clinically stable at the Week 1 study visit, the dose of LDMTX was increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose of LDMTX was increased to 15 mg once a week through Week 24. Participants who did not meet the criteria for dose escalation was re-evaluated at the following study visit. In addition to LDMTX, all participants also received 1 mg of folic acid once a day from study entry throughout Week 24. After taking the final dose of LDMTX, all participants continued taking folic acid for an additional 4 weeks.
  LDMTX: LDMTX 5 mg: one 5-mg capsule by mouth once weekly
  LDMTX 10 mg: two 5-mg capsules by mouth once weekly
  LDMTX 15 mg: three 5-mg capsules by mouth once weekly
  Folic acid: 1-mg tablet of folic acid by mouth once a day
- Placebo: From study entry through Week 1, participants received 5 mg of placebo once a week. For participants who were clinically stable at the Week 1 study visit, the dose of placebo was increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose of placebo was increased to 15 mg once a week through Week 24. Participants who did not meet the criteria for dose escalation was re-evaluated at the following study visit. In addition to placebo, all participants also received 1 mg of folic acid once a day from study entry throughout Week 24. After taking the final dose of placebo, all participants continued taking folic acid for an additional 4 weeks.
  Placebo: Placebo 5 mg: one 5-mg capsule by mouth once weekly
  Placebo 10 mg: two 5-mg capsules by mouth once weekly
  Placebo 15 mg: three 5-mg capsules by mouth once weekly
  Folic acid: 1-mg tablet of folic acid by mouth once a day
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 55 | 69
Percentage Change | -3.5 [-26.7 to 27.1] | 5.4 [-16.8 to 33.5]

9. Secondary Outcome: Percentage Change From Baseline to Week 24 in Interleukin-6 (IL-6)
Description: IL-6 is a marker of systemic inflammation. Change from baseline (Week 24 - baseline) was performed on the log10 scale and is thus presented as percentage change, i.e. (10^[fold-change] - 1) x 100%.
Time Frame: From Baseline to Week 24
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 59 | 70
Percentage Change | 13.4 [-1.3 to 30.3] | 21.3 [-0.2 to 47.4]

10. Secondary Outcome: Percentage Change From Baseline to Week 24 in Soluble CD 163 (sCD163)
Description: sCD163 is a marker of Macrophage activation. Change from baseline (Week 24 - baseline) was performed on the log10 scale and is thus presented as percentage change, i.e. (10^[fold-change] - 1) x 100%.
Time Frame: From Baseline to Week 24
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 56 | 69
Percentage Change | 2.7 [-4.2 to 10.1] | 7.5 [0.6 to 15.0]

11. Secondary Outcome: Percentage Change From Baseline to Week 24 in D-Dimer
Description: D-dimer (or D dimer) is a marker of coagulation activation. Change from baseline (Week 24 - baseline) was performed on the log10 scale and is thus presented as percentage change, i.e. (10^[fold-change] - 1) x 100%.
Time Frame: From Baseline to Week 24
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 56 | 69
Percentage Change | -1.5 [-10.6 to 8.5] | 9.9 [-3.3 to 24.9]

12. Secondary Outcome: Absolute Change From Baseline to Week 24 in Monocyte Levels
Description: Three categories of monocyte levels are presented: classical (CD14+CD16-), intermediate (CD14+CD16+), and non-classical (CD14dimCD16+). Absolute change from baseline (Week 24 - baseline) was analyzed on the measured scale, which is the percent of parent cells that express the subset of interest.
Time Frame: From Baseline to Week 24
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 56 | 68
Percent of Expression in Parent Cell
  Classical (CD14+CD16-) | -0.15 [-1.39 to 1.10] | 0.82 [-0.42 to 2.06]
  Intermediate (CD14+CD16+) | -0.07 [-0.77 to 0.62] | -0.51 [-1.32 to 0.29]
  Non-classical (CD14dimCD16+) | 0.21 [-0.66 to 1.08] | -0.29 [-0.89 to 0.31]

13. Secondary Outcome: Absolute Change From Baseline to Week 24 in Adhesion and Activation Indices
Description: The adhesion and activation indices of interest are the percentages of CD38+HLADR+ expressions in both parent CD4+ and CD8+ T cells. Absolute change from baseline (Week 24 - baseline) was analyzed on the measured scale, which is the percent of parent cells (either CD4+ or CD8+) that express CD38+HLADR+ cells.
Time Frame: From Baseline to Week 24
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 56 | 68
Percent of Expression in Parent Cell
  (CD3+CD4+) CD38+HLADR+ | -0.27 [-0.58 to 0.04] | 0.22 [-0.06 to 0.50]
  (CD3+CD8+) CD38+HLADR+ | -1.50 [-2.06 to -0.95] | 0.90 [-0.35 to 2.15]

14. Secondary Outcome: Absolute Change From Baseline to Week 24 in Homing Molecule (CX3CR1+) Expression
Description: CX3CR1+ is a cellular marker of immune activation. The outcome measured is the percentages of CX3CR1+ expressions in both parent CD4+ and CD8+ T cells. Absolute change from baseline (Week 24 - baseline) was analyzed on the measured scale, which is the percent of parent cells (either CD4+ or CD8+) that express CX3CR1+ cells.
Time Frame: From Baseline to Week 24
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Percent of Expression in Parent Cell
Arm/Group | Low-dose Methotrexate (LDMTX) | Placebo
Number analyzed (Participants) | 56 | 68
Percent of Expression in Parent Cell
  (CD3+CD4+) CX3CR1+ | -0.30 [-0.80 to 0.20] | 0.03 [-0.55 to 0.60]
  (CD3+CD8+) CX3CR1+ | -0.83 [-2.76 to 1.11] | 0.39 [-1.13 to 1.92]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) reported from study enrollment until study completion at 36 weeks.
Description: All serious adverse events, all AEs that led to a change in treatment, all signs and symptoms grade 2 or higher, all laboratory abnormalities grade 3 or higher and any of following targeted medical conditions: cardiovascular, hematologic, infectious, and neoplastic diseases (including mycobacterial infections, thrush, oral ulcers); hepatobilary, lymphoproliferative, renal, and pulmonary disorders; CDC category C AIDS conditions, regardless of grade.
Groups:
- LDMTX: From study entry through Week 1, participants received either 5 mg of LDMTX once a week. For participants who were clinically stable at the Week 1 study visit, the dose of LDMTX was increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose of LDMTX was increased to 15 mg once a week through Week 24. Participants who did not meet the criteria for dose escalation was re-evaluated at the following study visit. In addition to LDMTX, all participants also received 1 mg of folic acid once a day from study entry throughout Week 24. After taking the final dose of LDMTX, all participants continued taking folic acid for an additional 4 weeks.
- Placebo: From study entry through Week 1, participants received either 5 mg of placebo once a week. For participants who were clinically stable at the Week 1 study visit, the dose of placebo was increased to 10 mg once a week through Week 12. For participants who were clinically stable at the Week 12 study visit, the dose of placebo was increased to 15 mg once a week through Week 24. Participants who did not meet the criteria for dose escalation was re-evaluated at the following study visit. In addition to placebo, all participants also received 1 mg of folic acid once a day from study entry throughout Week 24. After taking the final dose of placebo, all participants continued taking folic acid for an additional 4 weeks.
Arm/Group | LDMTX | Placebo
All-Cause Mortality (participants affected / at risk) | 2/86 | 0/90
Serious Adverse Events (participants affected / at risk) | 9/86 | 8/90
Other Adverse Events (participants affected / at risk) | 81/86 | 76/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDMTX (N=86) | Placebo (N=90)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis shigella (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDMTX (N=86) | Placebo (N=90)
Nausea (Gastrointestinal disorders) | 5 | 2
Fatigue (General disorders) | 8 | 6
Malaise (General disorders) | 2 | 6
Pyrexia (General disorders) | 5 | 6
Alanine aminotransferase increased (Investigations) | 10 | 11
Aspartate aminotransferase increased (Investigations) | 11 | 15
Blood alkaline phosphatase increased (Investigations) | 3 | 6
Blood bicarbonate decreased (Investigations) | 12 | 9
Blood bilirubin increased (Investigations) | 12 | 11
Blood cholesterol increased (Investigations) | 37 | 27
Blood creatinine increased (Investigations) | 19 | 12
Blood glucose decreased (Investigations) | 12 | 3
Blood glucose increased (Investigations) | 38 | 39
Blood potassium decreased (Investigations) | 5 | 6
Blood sodium decreased (Investigations) | 19 | 14
Low density lipoprotein increased (Investigations) | 21 | 14
Neutrophil count decreased (Investigations) | 7 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No